CLINICAL TRIAL: NCT01565590
Title: Effects of Dexmedetomidine on Inflammatory Cytokines in Patients With Aneurysmal Subarachnoid Hemorrhage
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow enrollment along with new competing studies, investigators decided to stop study
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Shaun Keegan, Clinical Pharmacy Specialist, Critical Care, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-11-22-01
Record Dates: First submitted 2012-03-23; First posted 2012-03-28 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal
Keywords: aneurysmal subarachnoid hemorrhage; dexmedetomidine; cytokines
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propofol (Active Comparator)
  Interventions: Drug: propofol
- Dexmedetomidine (Experimental)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — 0.2-1.5 mcg/kg/hr
  Arms: Dexmedetomidine
Drug: propofol — 5-80 mcg/kg/min
  Arms: Propofol

SUMMARY:
The purpose of this research is to compare patients with aneurysmal subarachnoid hemorrhage on dexmedetomidine compared to propofol to assess if one group has decreased inflammation. The investigators hypothesis is that the group assigned to receive dexmedetomidine will have a more profound decrease in markers of inflammation over time.

ELIGIBILITY:
Inclusion Criteria:

* Aneurysmal subarachnoid hemorrhage
* World Federation of Neurological Surgeons (WFNS) grade 4-5 (see table below)
* Surgical intervention with clip or coil
* Placement of cerebrospinal fluid drain (lumbar or ventricular)
* Mechanically ventilated at start of infusion

Exclusion Criteria:

* Hemodynamic instability (SBP < 100, HR <60, or on continuous infusion of catecholamines) at screening
* Heart failure class III or IV (New York Heart Association)
* Renal failure (RIFLE classification - see table below)
* Liver failure (serum protein < 3 g/dL and total bilirubin > 5 mg/dL)
* Known or suspected brain death
* Pregnancy
* Unable to receive dexmedetomidine within 48 hours of injury and 4 hours of surgery
* Allergy to dexmedetomidine
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Changes between serum and CSF cytokines over 48 hours | 0, 24 and 48 hours
  Measure the baseline level (at enrollment) of inflammatory markers tumor necrosis factor-alpha (TNF-α), interleukin-6 (IL-6), glial fibrially acidic protein (GFAP), and malondialdehyde (MDA) as measured in both serum and cerebrospinal fluid (CSF) in 10 patients with aneurysmal subarachnoid hemorrhage (aSAH).

SECONDARY OUTCOMES:
Sedative and analgesic medication requirements | 2 weeks
  Sedation requirements between the two groups will be assessed by comparing total daily dose and average daily fentanyl doses in the 24 hours following surgery. The total number of patients requiring propofol rescue in the dexmedetomidine group and the total daily dose and average daily dose of the propofol used in the dexmedetomidine group will be recorded.
Sedation scores (RASS and CAM-ICU) | 2 weeks
ICU length of stay | 2 weeks
Hospital length of stay | 2 weeks
Glasgow Outcome Scores Extended (GOSE) at discharge | 2 weeks
Incidence of delayed cerebral ischemia (DCI) | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Cincinnati, Ohio, United States